CLINICAL TRIAL: NCT06532240
Title: Initiation of Methylene Blue for Septic Shock in Adults: A Randomized Clinical Trial
Brief Title: Methylene Blue for the Treatment of Septic Shock
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Qing-quan Lv, Principal Investigator, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024ky202
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Septic Shock
Keywords: septic shock; methylene blue; mortality
MeSH Terms: conditions — Shock, Septic | interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylene Blue (Experimental): Methylene Blue 100mg will be diluted in 40ml 5% dextrose solution. Methylene Blue(1 mg/kg/IBW iv over 30min+0.25mg/kg/h x 6h) x 5-days/ discontinution of norepinephrine /ICU discharge (whichever occurred first).
  Interventions: Drug: Methylene Blue
- Placebo (Placebo Comparator): 5% dextrose solution in a volume to match experimental arm component.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylene Blue — Methylene Blue 100mg will be diluted in 40ml 5% dextrose solution.The patient will receive Methylene Blue bolus with a dose of 1 mg/kg (Ideal Body Weight) over 30 minutes,followed by 0.25mg/kg/h as a continuous infusion for 6 hours for 5 days or discontinution of norepinephrine or until ICU discharge, whichever occurred first.
  Other Names: MB
  Arms: Methylene Blue
Drug: Placebo — An identical volume of 5% dextrose solution from the placebo drug bag will be administered to patients using the same protocol as intervention arm.
  Other Names: 5%GS
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of methylene blue among adult patients with septic shock.

DETAILED DESCRIPTION:
Septic Shock is a leading cause of morbidity and mortality in critically ill patients worldwide.

A potential benefit of methylene blue in the treatment of septic shock has recently been described by Estrada. In patients with septic shock, methylene blue initiated within 24 h reduced time to vasopressor discontinuation and increased vasopressor-free days at 28 days. It also reduced length of stay in ICU and hospital without adverse effects.

In this randomized controlled trial, we aim to evaluate the efficacy and safety of methylene blue on septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years old or older;
2. diagnosis of septic shock within 12 h.

Exclusion Criteria:

1. recent intake (4-weeks) of selective serotonin re-uptake inhibitors;
2. pregnant;
3. definitive pulmonary hypertension or chronic pulmonary heart disease;
4. known glucose-6 phosphate dehydrogenase (G-6PD) deficiency;
5. known allergy to methylene blue, phenothiazines, or food dyes;
6. anticipated death from a preexisting disease within 90 days after randomization (as determined by the enrolling physician);
7. refusal of the attending staff or patient family;
8. participated in other study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Time to shock reversal | 90 days after randomization
  Time to shock reversal was defined as the time from randomization to shock reversal.Reversal of shock was defined as the maintenance of a systolic blood pressure of at least 90 mmHg without vasopressor support for at least 24 h.

SECONDARY OUTCOMES:
28-day mortality | 28 days after randomization
  All-cause mortality at day 28 after randomization
90-day mortality | 90 days after randomization
  All-cause mortality at day 90 after randomization
ICU mortality | 90 days after randomization
  All-cause mortality at ICU discharge
Hospital mortality | 90 days after randomization
  All-cause mortality at hospital discharge

OTHER OUTCOMES:
ICU length of stay | 90 days after randomization
  Time in days until ICU discharge
hospital length of stay | 90 days after randomization
  Time in days until hospital discharge
ICU-free days up to day 28 | 28 days after randomization
  Total number of days alive and free of ICU stay during the 28 days after randomization.
vasopressor-free days up to day 28 | 28 days after randomization
  Total number of days alive and free of vasopressor during the 28 days after randomization.
ventilator support-free days up to day 28 | 28 days after randomization
  Total number of days alive and free of ventilator support during the 28 days after randomization.
CRRT-free days up to day 28 | 28 days after randomization
  Total number of days alive and free of CRRT during the 28 days after randomization.
72h lactate | 72 hours after randomization
  lactate level at 72h after randomization
72h Delta SOFA | 72 hours after randomization
  Initial SOFA score at enrollment-SOFA score after 72 h;If the patient discharged within 72 h after being enrolled in the study, the SOFA score at discharge was used for the analysis.
72h P/F | 72 hours after randomization
  P/F at 72h after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Qingquan Lyu, Master, Principal Investigator — Northern Jiangsu People's Hospital
Locations (1):
- Northern Jiangsu people's hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No